CLINICAL TRIAL: NCT01769469
Title: Renal, Endocrine, and Bone Changes in Response to Treatment With Coformulated Emtricitabine-Tenofovir for Pre-Exposure HIV Prophylaxis (PrEP) in HIV Uninfected Young Men Who Have Sex With Men.
Brief Title: Renal, Endocrine, and Bone Changes in Response to FTC/TDF in Uninfected Young Men Who Have Sex With Men (YMSM).
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: ATN 117 Version 2.0
Record Dates: First submitted 2013-01-14; First posted 2013-01-16 (Estimated); Results first posted 2019-03-11 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2018-11

CONDITIONS: HIV Infection
Keywords: Tenofovir; Emtricitabine; Truvada; Renal, endocrine, bone changes; HIV prevention; PrEP
MeSH Terms: conditions — HIV Infections | interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and urine samples to measure: Calcium-Phosphate Balance, Bone Turnover, Renal Glomerular Function, Renal Tubular Function.
  Dried blood spots (DBS) for FTC and Tenofovir (TFV)concentrations; red blood cell (RBC) for TFV-diphosphate (DP); plasma for FTC, TFV; peripheral blood mononuclear cells (PBMC) for TFV-DP and FTC-triphosphate (TP) collected as part of ATN 110 and ATN 113 will be used in the ATN 117 analysis.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subjects Enrolled in ATN 110 or ATN 113: A subset of 100 participants who are enrolled in the ATN 110 or ATN 113 study will be recruited for participation in this study. There is no treatment or intervention for this study; however, all subjects will be on daily coformulated tenofovir/emtricitabine (TDF/FTC (Truvada®)) as part of the ATN 110 or ATN 113 study.
  Interventions: Drug: FTC/TDF (Truvada®)

INTERVENTIONS:
Drug: FTC/TDF (Truvada®) — There are no interventions for this study except that subjects will be administered FTC/TDF (Truvada®) will be administered as part of ATN 110 and ATN 113.
  Other Names: Truvada®

SUMMARY:
This is a prospective observational cohort sub-study of subjects enrolled in the Adolescent Medicine Trials Network for HIV/AIDS Interventions (ATN) 110 (NCT01772823) or ATN 113 (NCT01769456), which is a prospective interventional trial.

DETAILED DESCRIPTION:
This is a prospective observational cohort sub-study of subjects enrolled in the ATN 110 (NCT01772823) or ATN 113 (NCT01769456) study. All subjects will be followed for at least 48 weeks. Subjects who meet specific bone or renal criteria at Week 48 of the ATN 110 (NCT01772823) or ATN 113 (NCT01769456) study will be followed for an additional 48 weeks in the Extension Phase of ATN 110 (NCT01772823) or ATN 113 (NCT01769456) and ATN 117 (NCT01769469). The maximum duration of participation will be 96 weeks.

There is no therapeutic intervention specific to this sub-study, and there are no extra study visits required for participation in this sub-study. Questionnaires will be administered and blood and urine samples for laboratory evaluation of potential emtricitabine (FTC)/tenofovir (TDF) (Truvada®) toxicities will be obtained for this sub-study at visits that are required by the ATN 110 (NCT01772823) or ATN 113 (NCT01769456) study. Measurement of bone mineral density (BMD) and bone mineral content (BMC) by dual-energy X-ray absorptiometry (DXA) scan are planned as a part of the ATN 110 (NCT01772823) and ATN 113 (NCT01769456) studies, and results will be utilized for the analysis in this study. This study does not require extra BMD or BMC measurements.

ELIGIBILITY:
Inclusion Criteria:

* Has been enrolled in ATN 110 (NCT01772823) or ATN 113 (NCT01769456) , and
* Willing and able to provide written informed consent

Exclusion Criteria:

-Subjects exempted from undergoing DXA scans in ATN 110 (NCT01772823) or ATN 113 (NCT01769456) are not eligible to enroll in ATN 117 (NCT01769469).

Ages: 15 Years to 22 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Individuals between the ages 15 years 0 days to 22 years 364 days, who are enrolled in ATN 110 (NCT01772823) or ATN 113 (NCT01769456) , and agree to enter this sub-study at the same time they begin ATN 110 or ATN 113.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2012-11; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Havens, MD, Study Chair — MACC Fund Research Center
Locations (12):
- United States (12):
  - Children's Hopsital of Los Angeles, Los Angeles, California
  - Children's Hospital of Denver, Aurora, Colorado
  - University of Miami, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Stroger Hospital and the CORE Center, Chicago, Illinois
  - Tulane University, New Orleans, Louisiana
  - Johns Hopkins University, Baltimore, Maryland
  - Fenway Institute, Boston, Massachusetts
  - Wayne State University, Detroit, Michigan
  - Children's Hopsital of Philadelphia, Philadelphia, Pennsylvania
  - St. Jude Childrens Research Hospital, Memphis, Tennessee
  - Baylor College of Medicine, Houston, Texas

REFERENCES:
- [Result] Havens PL, Stephensen CB, Van Loan MD, Schuster GU, Woodhouse LR, Flynn PM, Gordon CM, Pan CG, Rutledge B, Liu N, Wilson CM, Hazra R, Hosek SG, Anderson PL, Seifert SM, Kapogiannis BG, Mulligan K; Adolescent Medicine Trials Network for HIV/AIDS Interventions 117 study team. Decline in Bone Mass With Tenofovir Disoproxil Fumarate/Emtricitabine Is Associated With Hormonal Changes in the Absence of Renal Impairment When Used by HIV-Uninfected Adolescent Boys and Young Men for HIV Preexposure Prophylaxis. Clin Infect Dis. 2017 Feb 1;64(3):317-325. doi: 10.1093/cid/ciw765. Epub 2016 Nov 15. PMID 28013265
- [Derived] Havens PL, Tamhane A, Stephensen CB, Schuster GU, Gordon CM, Liu N, Wilson CM, Hosek SG, Anderson PL, Kapogiannis BG, Mulligan K. Short Communication: Association of Vitamin D Insufficiency and Protective Tenofovir Diphosphate Concentrations with Bone Toxicity in Adolescent Boys and Young Men Using Tenofovir Disoproxil Fumarate/Emtricitabine for HIV Pre-Exposure Prophylaxis. AIDS Res Hum Retroviruses. 2019 Feb;35(2):123-128. doi: 10.1089/AID.2018.0096. Epub 2018 Nov 5. PMID 30280906
- [Derived] Havens PL, Long D, Schuster GU, Gordon CM, Price G, Wilson CM, Kapogiannis BG, Mulligan K, Stephensen CB; Adolescent Medicine Trials Network for HIV/AIDS Interventions (ATN) 117 and 109 study teams. Tenofovir disoproxil fumarate appears to disrupt the relationship of vitamin D and parathyroid hormone. Antivir Ther. 2018;23(7):623-628. doi: 10.3851/IMP3269. Epub 2018 Sep 27. PMID 30260797
- See also: ATN Website — http://www.atnonline.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The research was conducted at 11 clinical sites. Accrual was open between November 2012 and December 2013.
Groups:
- Subjects Enrolled in ATN 110 or ATN 113: A subset of 101 participants who are enrolled in the ATN 110 or ATN 113 study will be recruited for participation in this study. There is no treatment or intervention for this study; however, all subjects will be on daily coformulated tenofovir (TDF)/emtricitabine (FTC) (TDF/FTC (Truvada®)) as part of the ATN 110 or ATN 113 study.
  FTC/TDF (Truvada®): There are no interventions for this study except that subjects will be administered FTC/TDF (Truvada®) will be administered as part of ATN 110 and ATN 113.
Period: Overall Study
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Started | 101
Completed | 66
Not Completed | 35
Not completed — Consent Withdrawn | 5
Not completed — Moved Out Of Area | 3
Not completed — Lost to Follow-up | 17
Not completed — Prem D/C from ATN 110/113 For Any Reason | 7
Not completed — Subject Confirmed HIV Positive | 3

BASELINE CHARACTERISTICS:
Groups:
- Subjects Enrolled in ATN 110 or ATN 113: A subset of 101 participants who are enrolled in the ATN 110 or ATN 113 study will be recruited for participation in this study. There is no treatment or intervention for this study; however, all subjects will be on daily coformulated tenofovir/emtricitabine (TDF/FTC (Truvada®)) as part of the ATN 110 or ATN 113 study.
  FTC/TDF (Truvada®): There are no interventions for this study except that subjects will be administered FTC/TDF (Truvada®) will be administered as part of ATN 110 and ATN 113.
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.62 (1.80)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 101
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian/Pacific Islander | 2
  Black/African American | 43
  White | 16
  White/Hispanic | 14
  Other/Mixed Race | 26
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black/African American | 52
  Non-Black/African American | 49
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 34
  Non-Hispanic | 67
Parathyroid hormone (PTH) [Median (Full Range); unit: pg/mL] — Population: Subjects with available data
  pg/mL
    number analyzed (Participants) | 100
    (all) | 27.07 [10.44 to 84.26]
Fibroblast growth factor 23 (FGF23) [Median (Full Range); unit: pg/mL] — Population: Subjects with available data
  pg/mL
    number analyzed (Participants) | 100
    (all) | 38.78 [16.92 to 123.81]
1,25-dihydroxy vitamin D (1,25-OHD RIA) [Median (Full Range); unit: pmol/L] — Population: Subjects with available data
  pmol/L
    number analyzed (Participants) | 100
    (all) | 160.71 [61.88 to 343.63]
Tubular reabsorption of phosphate (TRP) [Median (Full Range); unit: % (of filtered phosphorus reabsorbed)] | 91.40 [66.32 to 99.91]
Actual Free 123(OH)D [Median (Full Range); unit: fmol/L] — Population: Subjects with available data
  fmol/L
    number analyzed (Participants) | 100
    (all) | 994.88 [250.21 to 4176.15]
Estimated glomerular filtration rate (eGFR) [Median (Full Range); unit: mL/min/1.73^2] | 127.50 [70.74 to 280.61]
Serum Creatinine (SCr) [Median (Full Range); unit: mg/dL] | 0.86 [0.61 to 1.29]
Serum Calcium (SCa) [Median (Full Range); unit: mg/dL] | 9.80 [8.62 to 10.98]
Urinary Calcium/ Urinary Creatinine ratio (UCa/UCr) [Median (Full Range); unit: ratio] | 0.06 [0.00 to 0.23]
Serum Phosphate (SPO4) [Median (Full Range); unit: mmol/L] | 1.16 [0.83 to 1.74]
Urine Glucose (UGluc) [Median (Full Range); unit: mg/dL] | 0.07 [0.01 to 0.19]
Urine retinol binding protein to urine creatinine ratio (URBP/UCr) [Median (Full Range); unit: mcg/g] — Population: Subjects with data available.
  mcg/g
    number analyzed (Participants) | 100
    (all) | 7092.50 [672.40 to 98673.09]
Urine beta-2 microglobulin (UB2MG) [Median (Full Range); unit: ng/mL] — Population: Subjects with available data
  ng/mL
    number analyzed (Participants) | 97
    (all) | 170.04 [9.78 to 3767.40]
Urine protein to urine creatinine ratio (UProt/UCr) [Median (Full Range); unit: ratio] | 0.05 [0.03 to 0.20]
Osteocalcin (OC) [Median (Full Range); unit: mcg/L] — Population: Subjects with available data
  mcg/L
    number analyzed (Participants) | 100
    (all) | 9.50 [1.03 to 17.31]
C-telopeptide (CTX) [Median (Full Range); unit: pg/mL] — Population: Subjects with available data
  pg/mL
    number analyzed (Participants) | 100
    (all) | 935.76 [278.54 to 2038.42]
Lumbar spine bone mineral density (BMD) [Median (Full Range); unit: g/cm^2] | 1.09 [0.76 to 1.49]
Femoral neck bone mineral density (BMD) [Median (Full Range); unit: g/cm^2] — Population: Subjects with available data
  g/cm^2
    number analyzed (Participants) | 100
    (all) | 1.03 [0.65 to 1.43]
Total body bone mineral content (BMC) [Median (Full Range); unit: g] | 2690.83 [1905.32 to 3702.70]

OUTCOME MEASURES:

1. Primary Outcome: Magnitude of Change (Fold Change) in Parathyroid Hormone (PTH) From Baseline to Week 48
Description: The magnitude of change in PTH will be measured between Baseline and Week 48. For any given variable, at a given time point, the magnitude of change is the fold change compared to the baseline value (if multiplied by 100 would be the percent change from baseline).
Time Frame: Baseline and Week (wk) 48
Population: Subjects with PTH data at baseline and Week 48
Measure: Median (Full Range); unit: fold change
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 70
fold change | 1.08 [0.61 to 2.59]

2. Secondary Outcome: Change in Renal-endocrine-bone Biochemistry and Pathophysiology: Fibroblast Growth Factor 23 (FGF23), Change From Baseline to Week 48
Time Frame: Baseline and wk 48
Population: Subjects with data for baseline and Week 48
Measure: Median (Full Range); unit: pg/ML
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 70
pg/ML | -1.50 [-25.50 to 65.18]
Statistical Analysis 1: Comparison: Subjects Enrolled in ATN 110 or ATN 113; Test of difference at Week 48 from baseline; Test type: Other; p = 0.2085, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Change in Renal-endocrine-bone Biochemistry and Pathophysiology: Fibroblast Growth Factor 23 (FGF23), Magnitude of Fold Change
Description: The magnitude of change in FGF23 will be measured between Baseline and Week 48. For any given variable, at a given time point, the magnitude of change is the fold change compared to the baseline value (if multiplied by 100 would be the percent change from baseline).
Time Frame: Baseline and wk 48
Population: Subjects with data for baseline and Week 48
Measure: Median (Full Range); unit: fold change
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 70
fold change | 0.96 [0.54 to 2.47]

4. Secondary Outcome: Change in Renal-endocrine-bone Biochemistry and Pathophysiology: Fibroblast Growth Factor 23 (FGF23), Most Extreme Fold Change
Description: Most extreme fold change: This is the highest or lowest value measured as fold change from the baseline value of that variable.
Time Frame: Baseline, Weeks 4, 8, 12, 24, 36 and 48
Population: Subjects with at least two measurements available for comparison
Measure: Median (Full Range); unit: fold change
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 90
fold change | 1.18 [0.67 to 2.47]

5. Secondary Outcome: Change in Renal-endocrine-bone Biochemistry and Pathophysiology: Fibroblast Growth Factor 23 (FGF23), Time to Most Extreme Fold Change
Description: The time to most extreme fold change is the study week associated with the most extreme fold change or extreme percent change from baseline.
Time Frame: Baseline, Weeks 4, 8, 12, 24, 36, and 48
Population: Subjects with at least two measurements available for comparison
Measure: Median (Full Range); unit: weeks
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 90
weeks | 12.00 [4.00 to 48.00]

6. Secondary Outcome: Change in Renal-endocrine-bone Biochemistry and Pathophysiology: 1,25 Dihydroxy Vitamin D (1,25 OHD), Change From Baseline to Week 48
Time Frame: Baseline and wk 48
Population: Subjects with data for baseline and Week 48
Measure: Median (Full Range); unit: pmol/L
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 71
pmol/L | -8.61 [-135.40 to 197.62]
Statistical Analysis 1: Comparison: Subjects Enrolled in ATN 110 or ATN 113; Test type: Superiority; p = 0.2452, Wilcoxon Signed Rank Test

7. Secondary Outcome: Change in Renal-endocrine-bone Biochemistry and Pathophysiology: 1,25 OHD, Magnitude of Fold Change
Description: The magnitude of change in 1,25 OHD will be measured between Baseline and Week 48. For any given variable, at a given time point, the magnitude of change is the fold change compared to the baseline value (if multiplied by 100 would be the percent change from baseline).
Time Frame: Baseline and wk 48
Population: Subjects with data for baseline and Week 48
Measure: Median (Full Range); unit: fold change
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 71
fold change | 0.95 [0.42 to 2.87]

8. Secondary Outcome: Change in Renal-endocrine-bone Biochemistry and Pathophysiology: 1,25 OHD, Most Extreme Fold Change
Description: as for outcome 4
Time Frame: Baseline, Weeks 4, 8, 12, 24, 36 and 48
Population: Subjects with at least two measurements available for comparison
Measure: Median (Full Range); unit: fold change
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 90
fold change | 1.33 [0.74 to 3.06]

9. Secondary Outcome: Change in Renal-endocrine-bone Biochemistry and Pathophysiology: 1,25 OHD, Time to Most Extreme Fold Change
Description: as for outcome 5
Time Frame: Baseline, Weeks 4, 8, 12, 24, 36, and 48
Population: Subjects with at least two measurements available for comparison
Measure: Median (Full Range); unit: weeks
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 90
weeks | 12.00 [4.00 to 48.00]

10. Secondary Outcome: Change in Renal-endocrine-bone Biochemistry and Pathophysiology: Tubular Reabsorption of Phosphate (TRP), Change From Baseline to Week 48
Time Frame: Baseline and wk 48
Population: Subjects with data for baseline and Week 48
Measure: Median (Full Range); unit: percentage of phosphorus reabsorbed
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 71
percentage of phosphorus reabsorbed | -0.57 [-10.80 to 10.54]

11. Secondary Outcome: Change in Renal-endocrine-bone Biochemistry and Pathophysiology: TRP, Magnitude of Fold Change
Description: The magnitude of change in TRP will be measured between Baseline and Week 48. For any given variable, at a given time point, the magnitude of change is the fold change compared to the baseline value (if multiplied by 100 would be the percent change from baseline).
Time Frame: Baseline and wk 48
Population: Subjects with data for baseline and Week 48
Measure: Median (Full Range); unit: fold change
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 71
fold change | 0.99 [0.89 to 1.13]

12. Secondary Outcome: Change in Renal-endocrine-bone Biochemistry and Pathophysiology: TRP, Most Extreme Fold Change
Description: as for outcome 4
Time Frame: Baseline, Weeks 4, 8, 12, 24, 36 and 48
Population: Subjects with at least two measurements available for comparison
Measure: Median (Full Range); unit: fold change
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 91
fold change | 1.05 [0.97 to 1.47]

13. Secondary Outcome: Change in Renal-endocrine-bone Biochemistry and Pathophysiology: TRP, Time to Most Extreme Fold Change
Description: as for outcome 5
Time Frame: Baseline, Weeks 4, 8, 12, 24, 36, and 48
Population: Subjects with at least two measurements available for comparison
Measure: Median (Full Range); unit: weeks
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 91
weeks | 24.00 [4.00 to 48.00]

14. Secondary Outcome: Change in Renal-endocrine-bone Biochemistry and Pathophysiology: Glomerular Filtration Rate (GFR), Change From Baseline to Week 48
Time Frame: Baseline and wk 48
Population: Subjects with data for baseline and Week 48
Measure: Median (Full Range); unit: ml/min/1.73m^2
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 70
ml/min/1.73m^2 | 3.06 [-32.03 to 95.42]
Statistical Analysis 1: Comparison: Subjects Enrolled in ATN 110 or ATN 113; Test type: Superiority; p = .0806, Wilcoxon Signed Rank Test

15. Secondary Outcome: Change in Renal-endocrine-bone Biochemistry and Pathophysiology: GFR, Magnitude of Fold Change
Description: The magnitude of change in GFR will be measured between Baseline and Week 48. For any given variable, at a given time point, the magnitude of change is the fold change compared to the baseline value (if multiplied by 100 would be the percent change from baseline).
Time Frame: Baseline and wk 48
Population: Subjects with data for baseline and Week 48
Measure: Median (Full Range); unit: fold change
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 70
fold change | 1.02 [0.76 to 1.83]

16. Secondary Outcome: Change in Renal-endocrine-bone Biochemistry and Pathophysiology: GFR, Most Extreme Fold Change
Description: as for outcome 4
Time Frame: Baseline, Weeks 4, 8, 12, 24, 36 and 48
Population: Subjects with at least two measurements available for comparison
Measure: Median (Full Range); unit: fold change
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 90
fold change | 1.10 [0.77 to 1.83]

17. Secondary Outcome: Change in Renal-endocrine-bone Biochemistry and Pathophysiology: GFR, Time to Most Extreme Fold Change
Description: as for outcome 5
Time Frame: Baseline, Weeks 4, 8, 12, 24, 36, and 48
Population: Subjects with at least two measurements available for comparison
Measure: Median (Full Range); unit: weeks
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 90
weeks | 24.00 [4.00 to 48.00]

18. Secondary Outcome: Change in Renal-endocrine-bone Biochemistry and Pathophysiology: PTH, Most Extreme Fold Change
Description: as for outcome 4
Time Frame: Baseline, Weeks 4, 8, 12, 24, 36 and 48
Population: Subjects with at least two measurements available for comparison
Measure: Median (Full Range); unit: fold change
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 90
fold change | 1.35 [0.59 to 2.81]

19. Secondary Outcome: Change in Renal-endocrine-bone Biochemistry and Pathophysiology: PTH, Time to Most Extreme Fold Change
Description: as for outcome 5
Time Frame: Baseline, Weeks 4, 8, 12, 24, 36, and 48
Population: Subjects with at least two measurements available for comparison
Measure: Median (Full Range); unit: weeks
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 90
weeks | 24.00 [4.00 to 48.00]

20. Secondary Outcome: Change in Renal-endocrine-bone Biochemistry and Pathophysiology: Serum Creatinine (SCr), Time to Most Extreme Fold Change
Description: as for outcome 5
Time Frame: Baseline, Weeks 4, 8, 12, 24, 36, and 48
Population: Subjects with at least two measurements available for comparison
Measure: Median (Full Range); unit: weeks
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 91
weeks | 8.00 [4.00 to 48.00]

21. Secondary Outcome: Change in Renal-endocrine-bone Biochemistry and Pathophysiology: PTH, Slope of the Curve of Baseline to Most Extreme Fold Change
Description: The slope from baseline to most extreme fold change can be expressed as:
  Slope = [(Most extreme fold change) * (baseline value) - (baseline value)] / [(Time to most extreme fold change) - (time of the baseline value)]
Time Frame: Baseline, Weeks 4, 8, 12, 24, 36, and 48
Population: Subjects with at least two measurements available for comparison
Measure: Median (Full Range); unit: (pg/mL)/ weeks
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 90
(pg/mL)/ weeks | 0.51 [-8.33 to 11.43]

22. Secondary Outcome: Change in Renal-endocrine-bone Biochemistry and Pathophysiology: FGF23, Slope of the Curve of Baseline to Most Extreme Fold Change
Description: as for outcome 21
Time Frame: Baseline, Weeks 4, 8, 12, 24, 36, and 48
Population: Subjects with at least two measurements available for comparison
Measure: Median (Full Range); unit: (pg/mL)/ weeks
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 90
(pg/mL)/ weeks | 0.39 [-5.14 to 9.21]

23. Secondary Outcome: Change in Renal-endocrine-bone Biochemistry and Pathophysiology: 1,25-OHD, Slope of the Curve of Baseline to Most Extreme Fold Change
Description: as for outcome 21
Time Frame: Baseline, Weeks 4, 8, 12, 24, 36, and 48
Population: Subjects with at least two measurements available for comparison
Measure: Median (Full Range); unit: (pmol/L)/ weeks
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 90
(pmol/L)/ weeks | 4.27 [-12.84 to 32.92]

24. Secondary Outcome: Change in Renal-endocrine-bone Biochemistry and Pathophysiology: TRP, Slope of the Curve of Baseline to Most Extreme Fold Change
Description: as for outcome 21
Time Frame: Baseline, Weeks 4, 8, 12, 24, 36, and 48
Population: Subjects with at least two measurements available for comparison
Measure: Median (Full Range); unit: (% phosphorus reabsorbed)/ weeks
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 91
(% phosphorus reabsorbed)/ weeks | 0.21 [-0.40 to 3.93]

25. Secondary Outcome: Change From Baseline to Week 48 in Serum Calcium (SCa)
Description: Serum calcium Week 48 difference from baseline
Time Frame: Baseline and wk 48
Population: Subjects with data for baseline and Week 48
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 70
mg/dL | -0.07 [-1.28 to 1.90]
Statistical Analysis 1: Comparison: Subjects Enrolled in ATN 110 or ATN 113; Test type: Other; p = 0.6545, Wilcoxon Signed Rank Test

26. Secondary Outcome: Magnitude of Most Extreme Fold Change: Serum Calcium (SCa)
Description: as for outcome 4
Time Frame: Baseline, Weeks 4, 8, 12, 24, 36, and 48
Population: Subjects with data available for at least two time points
Measure: Median (Full Range); unit: fold change
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 91
fold change | 1.03 [0.91 to 1.19]

27. Secondary Outcome: Time to Most Extreme Fold Change: Serum Calcium (SCa)
Description: as for outcome 5
Time Frame: Baseline, Weeks 4, 8, 12, 24, 36, and 48
Population: Subjects with at least two measurements available for comparison
Measure: Median (Full Range); unit: weeks
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 91
weeks | 12.00 [4.00 to 48.00]

28. Secondary Outcome: Slope of the Curve of Baseline to Most Extreme Fold Change: Serum Calcium (SCa)
Description: as for outcome 21
Time Frame: Baseline, Weeks 4, 8, 12, 24, 36, and 48
Population: Subjects with at least two measurements available for comparison
Measure: Median (Full Range); unit: (mg/dL)/ weeks
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 91
(mg/dL)/ weeks | 0.02 [-0.12 to 0.27]

29. Secondary Outcome: Change From Baseline to Week 48 in Urine Calcium (UCa) / Urine Creatinine (UCr)
Description: Urine Calcium (UCa) / Urine Creatinine (UCr) ratio Week 48 difference from baseline
Time Frame: Baseline and wk 48
Population: Subjects with data for baseline and Week 48
Measure: Median (Full Range); unit: ratio
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 71
ratio | 0.00 [-0.19 to 0.30]
Statistical Analysis 1: Comparison: Subjects Enrolled in ATN 110 or ATN 113; Test type: Other; p = 0.8739, Wilcoxon Signed Rank Test

30. Secondary Outcome: Magnitude of Most Extreme Fold Change: UCa/UCr Ratio
Description: as for outcome 4
Time Frame: Baseline, Weeks 4, 8, 12, 24, 36, and 48
Population: Subjects with at least two measurements available for comparison
Measure: Median (Full Range); unit: fold change
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 91
fold change | 1.95 [0.27 to 11.03]

31. Secondary Outcome: Time to Most Extreme Fold Change: UCa/UCr Ratio
Description: as for outcome 5
Time Frame: Baseline, Weeks 4, 8, 12, 24, 36, and 48
Population: Subjects with at least two measurements available for comparison
Measure: Median (Full Range); unit: weeks
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 91
weeks | 12.00 [4.00 to 48.00]

32. Secondary Outcome: Slope of the Curve of Baseline to Most Extreme Fold Change: UCa/UCr Ratio
Description: as for outcome 21
Time Frame: Baseline, Weeks 4, 8, 12, 24, 36, and 48
Population: Subjects with at least two measurements available for comparison
Measure: Median (Full Range); unit: (mg/mg)/ weeks
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 91
(mg/mg)/ weeks | 0.00 [-0.01 to 0.03]

33. Secondary Outcome: Change From Baseline to Week 48 in Serum Phosphate (SPO4)
Description: Serum Phosphate (SPO4) Week 48 difference from baseline
Time Frame: Baseline and wk 48
Population: Subjects with data for baseline and Week 48
Measure: Median (Full Range); unit: mmol/L
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 71
mmol/L | 0.00 [-0.67 to 0.47]

34. Secondary Outcome: Magnitude of Most Extreme Fold Change: SPO4
Description: as for outcome 4
Time Frame: Baseline, Weeks 4, 8, 12, 24, 36, and 48
Population: Subjects with at least two measurements available for comparison
Measure: Median (Full Range); unit: fold change
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 91
fold change | 1.14 [0.79 to 1.78]

35. Secondary Outcome: Time to Most Extreme Fold Change: SPO4
Description: as for outcome 5
Time Frame: Baseline, Weeks 4, 8, 12, 24, 36, and 48
Population: Subjects with at least two measurements available for comparison
Measure: Median (Full Range); unit: weeks
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 91
weeks | 12.00 [4.00 to 48.00]

36. Secondary Outcome: Slope of the Curve of Baseline to Most Extreme Fold Change: SPO4
Description: as for outcome 21
Time Frame: Baseline, Weeks 4, 8, 12, 24, 36, and 48
Population: Subjects with at least two measurements available for comparison
Measure: Median (Full Range); unit: (mmol/L)/ weeks
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 91
(mmol/L)/ weeks | 0.01 [-0.05 to 0.09]

37. Secondary Outcome: Change in Glomerular and Renal Tubular Function: Change From Baseline to Week 48 in Urine Retinol Binding Protein (URBP)/ Urine Creatinine (UCr)
Description: URBP/UCr Week 48 difference from baseline
Time Frame: Baseline and wk 48
Population: Subjects with data for baseline and Week 48
Measure: Median (Full Range); unit: mcg/g
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 69
mcg/g | -601.14 [-29433.03 to 42595.81]
Statistical Analysis 1: Comparison: Subjects Enrolled in ATN 110 or ATN 113; Test type: Other; p = 0.5014, Wilcoxon Signed Rank Test

38. Secondary Outcome: Change in Glomerular and Renal Tubular Function: Change From Baseline to Week 48 in Urine Beta-2 Microglobulin (UB2MG)
Description: UB2MG Week 48 difference from baseline
Time Frame: Baseline and wk 48
Population: Subjects with data for baseline and Week 48
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 67
ng/mL | -34.78 [-1252.73 to 597.59]
Statistical Analysis 1: Comparison: Subjects Enrolled in ATN 110 or ATN 113; Test type: Other; p = 0.2431, Wilcoxon Signed Rank Test

39. Secondary Outcome: Change in Glomerular and Renal Tubular Function: Change From Baseline to Week 48 in Urine Protein (UProt) / Urine Creatinine (UCr)
Description: UProt/ UCr Week 48 difference from baseline
Time Frame: Baseline and wk 48
Population: Subjects with data for baseline and Week 48
Measure: Median (Full Range); unit: ratio
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 71
ratio | 0.00 [-0.07 to 0.06]
Statistical Analysis 1: Comparison: Subjects Enrolled in ATN 110 or ATN 113; Test type: Other; p = 0.7209, Wilcoxon Signed Rank Test

40. Secondary Outcome: Change in Glomerular and Renal Tubular Function: Change From Baseline to Week 48 in Urine Glucose (UGluc)
Description: UGluc Week 48 difference from baseline
Time Frame: Baseline and wk 48
Population: Subjects with data for baseline and Week 48
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 71
mg/dL | -0.01 [-0.10 to 0.11]
Statistical Analysis 1: Comparison: Subjects Enrolled in ATN 110 or ATN 113; Test type: Other; p = 0.5379, Wilcoxon Signed Rank Test

41. Secondary Outcome: Change in Glomerular and Renal Tubular Function: Change From Baseline to Week 48 in Serum Creatinine (SCr)
Description: SCr Week 48 difference from baseline
Time Frame: Baseline and wk 48
Population: Subjects with data for baseline and Week 48
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 71
mg/dL | -0.01 [-0.12 to 0.27]
Statistical Analysis 1: Comparison: Subjects Enrolled in ATN 110 or ATN 113; Test type: Other; p = 0.7986, Wilcoxon Signed Rank Test

42. Secondary Outcome: Change in Glomerular and Renal Tubular Function: Magnitude of Fold Change at Week 48 in Urine Retinol Binding Protein (URBP)/ Urine Creatinine (UCr)
Description: The magnitude of change in URBP/UCr will be measured between Baseline and Week 48. For any given variable, at a given time point, the magnitude of change is the fold change compared to the baseline value (if multiplied by 100 would be the percent change from baseline).
Time Frame: Baseline and wk 48
Population: Subjects with data for baseline and Week 48
Measure: Median (Full Range); unit: fold change
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 69
fold change | 0.81 [0.00 to 11.94]

43. Secondary Outcome: Change in Glomerular and Renal Tubular Function: Magnitude of Fold Change at Week 48 in Urine Beta-2 Microglobulin (UB2MG)
Description: The magnitude of change in UB2MG will be measured between Baseline and Week 48. For any given variable, at a given time point, the magnitude of change is the fold change compared to the baseline value (if multiplied by 100 would be the percent change from baseline).
Time Frame: Baseline and wk 48
Population: Subjects with data for baseline and Week 48
Measure: Median (Full Range); unit: fold change
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 67
fold change | 0.72 [0.08 to 50.50]

44. Secondary Outcome: Change in Glomerular and Renal Tubular Function: Magnitude of Fold Change at Week 48 in Urine Protein (UProt)/ Urine Creatinine (UCr)
Description: The magnitude of change in UProt/UCr will be measured between Baseline and Week 48. For any given variable, at a given time point, the magnitude of change is the fold change compared to the baseline value (if multiplied by 100 would be the percent change from baseline).
Time Frame: Baseline and wk 48
Population: Subjects with data for baseline and Week 48
Measure: Median (Full Range); unit: fold change
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 71
fold change | 1.01 [0.43 to 2.17]

45. Secondary Outcome: Change in Glomerular and Renal Tubular Function: Magnitude of Fold Change at Week 48 in Urine Glucose (UGluc)
Description: The magnitude of change in UGluc will be measured between Baseline and Week 48. For any given variable, at a given time point, the magnitude of change is the fold change compared to the baseline value (if multiplied by 100 would be the percent change from baseline).
Time Frame: Baseline and wk 48
Population: Subjects with data for baseline and Week 48
Measure: Median (Full Range); unit: fold change
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 71
fold change | 0.94 [0.08 to 4.45]

46. Secondary Outcome: Change in Glomerular and Renal Tubular Function: Magnitude of Fold Change at Week 48 in Serum Creatinine (SCr)
Description: The magnitude of change in SCr will be measured between Baseline and Week 48. For any given variable, at a given time point, the magnitude of change is the fold change compared to the baseline value (if multiplied by 100 would be the percent change from baseline).
Time Frame: Baseline and wk 48
Population: Subjects with data for baseline and Week 48
Measure: Median (Full Range); unit: fold change
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 71
fold change | 0.99 [0.85 to 1.27]

47. Secondary Outcome: Change in Glomerular and Renal Tubular Function: Most Extreme Fold Change in Urine Retinol Binding Protein (URBP)/ Urine Creatinine (UCr)
Description: as for outcome 4
Time Frame: Baseline, Weeks 4, 8, 12, 24, 36 and 48
Population: Subjects with at least two measurements available for comparison
Measure: Median (Full Range); unit: fold change
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 90
fold change | 1.80 [0.44 to 15.27]

48. Secondary Outcome: Change in Glomerular and Renal Tubular Function: Most Extreme Fold Change in UB2MG
Description: as for outcome 4
Time Frame: Baseline, Weeks 4, 8, 12, 24, 36 and 48
Population: Subjects with at least two measurements available for comparison
Measure: Median (Full Range); unit: fold change
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 87
fold change | 2.59 [0.11 to 239.26]

49. Secondary Outcome: Change in Glomerular and Renal Tubular Function: Most Extreme Fold Change in UProt/UCr
Description: as for outcome 4
Time Frame: Baseline, Weeks 4, 8, 12, 24, 36 and 48
Population: Subjects with at least two measurements available for comparison
Measure: Median (Full Range); unit: fold change
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 91
fold change | 1.36 [0.42 to 4.46]

50. Secondary Outcome: Change in Glomerular and Renal Tubular Function: Most Extreme Fold Change in UGluc
Description: as for outcome 4
Time Frame: Baseline, Weeks 4, 8, 12, 24, 36 and 48
Population: Subjects with at least two measurements available for comparison
Measure: Median (Full Range); unit: fold change
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 91
fold change | 1.56 [0.62 to 11.34]

51. Secondary Outcome: Change in Glomerular and Renal Tubular Function: Most Extreme Fold Change in SCr
Description: as for outcome 4
Time Frame: Baseline, Weeks 4, 8, 12, 24, 36 and 48
Population: Subjects with at least two measurements available for comparison
Measure: Median (Full Range); unit: fold change
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 91
fold change | 1.09 [0.89 to 1.34]

52. Secondary Outcome: Change in Glomerular and Renal Tubular Function: Time to Most Extreme Fold Change in Urine Retinol Binding Protein (URBP)/ Urine Creatinine (UCr)
Description: as for outcome 5
Time Frame: Baseline, Weeks 4, 8, 12, 24, 36, and 48
Population: Subjects with at least two measurements available for comparison
Measure: Median (Full Range); unit: weeks
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 90
weeks | 12.00 [4.00 to 48.00]

53. Secondary Outcome: Change in Glomerular and Renal Tubular Function: Time to Most Extreme Fold Change in UB2MG
Description: as for outcome 5
Time Frame: Baseline, Weeks 4, 8, 12, 24, 36, and 48
Population: Subjects with at least two measurements available for comparison
Measure: Median (Full Range); unit: weeks
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 87
weeks | 12.00 [4.00 to 48.00]

54. Secondary Outcome: Change in Glomerular and Renal Tubular Function: Time to Most Extreme Fold Change in UProt/UCr
Description: as for outcome 5
Time Frame: Baseline, Weeks 4, 8, 12, 24, 36, and 48
Population: Subjects with at least two measurements available for comparison
Measure: Median (Full Range); unit: weeks
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 91
weeks | 24.00 [4.00 to 48.00]

55. Secondary Outcome: Change in Glomerular and Renal Tubular Function: Time to Most Extreme Fold Change in UGluc
Description: as for outcome 5
Time Frame: Baseline, Weeks 4, 8, 12, 24, 36, and 48
Population: Subjects with at least two measurements available for comparison
Measure: Median (Full Range); unit: weeks
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 91
weeks | 24.00 [4.00 to 48.00]

56. Secondary Outcome: Change in Glomerular and Renal Tubular Function: Slope of the Curve of Baseline to Most Extreme Fold Change in Urine Retinol Binding Protein (URBP)/ Urine Creatinine (UCr)
Description: as for outcome 21
Time Frame: Baseline, Weeks 4, 8, 12, 24, 36, and 48
Population: Subjects with at least two measurements available for comparison
Measure: Median (Full Range); unit: (mcg/g)/ weeks
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 90
(mcg/g)/ weeks | 270.70 [-742.00 to 6995.69]

57. Secondary Outcome: Change in Glomerular and Renal Tubular Function: Slope of the Curve of Baseline to Most Extreme Fold Change in UB2MG
Description: as for outcome 21
Time Frame: Baseline, Weeks 4, 8, 12, 24, 36, and 48
Population: Subjects with at least two measurements available for comparison
Measure: Median (Full Range); unit: (ng/mL)/ weeks
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 87
(ng/mL)/ weeks | 12.45 [-837.01 to 297.28]

58. Secondary Outcome: Change in Glomerular and Renal Tubular Function: Slope of the Curve of Baseline to Most Extreme Fold Change in UProt/UCr
Description: as for outcome 21
Time Frame: Baseline, Weeks 4, 8, 12, 24, 36, and 48
Population: Subjects with at least two measurements available for comparison
Measure: Median (Full Range); unit: Weeks^-1
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 91
Weeks^-1 | 0.00 [-0.01 to 0.03]

59. Secondary Outcome: Change in Glomerular and Renal Tubular Function: Slope of the Curve of Baseline to Most Extreme Fold Change in UGluc
Description: as for outcome 21
Time Frame: Baseline, Weeks 4, 8, 12, 24, 36, and 48
Population: Subjects with at least two measurements available for comparison
Measure: Median (Full Range); unit: (mg/dL)/ weeks
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 91
(mg/dL)/ weeks | 0.00 [-0.01 to 0.02]

60. Secondary Outcome: Change in Glomerular and Renal Tubular Function: Slope of the Curve of Baseline to Most Extreme Fold Change in Scr
Description: as for outcome 21
Time Frame: Baseline, Weeks 4, 8, 12, 24, 36, and 48
Population: Subjects with at least two measurements available for comparison
Measure: Median (Full Range); unit: (mg/dL)/ weeks
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 91
(mg/dL)/ weeks | 0.01 [-0.03 to 0.06]

61. Secondary Outcome: Change in Renal-endocrine-bone Biochemistry and Pathophysiology: Change From Baseline to Week 48 in Osteocalcin (OC)
Description: OC Week 48 difference from baseline
Time Frame: Baseline and wk 48
Population: Subjects with data for baseline and Week 48
Measure: Median (Full Range); unit: mcg/L
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 70
mcg/L | 0.05 [-6.17 to 7.77]
Statistical Analysis 1: Comparison: Subjects Enrolled in ATN 110 or ATN 113; Test type: Other; p = 0.8507, Wilcoxon Signed Rank Test

62. Secondary Outcome: Change in Renal-endocrine-bone Biochemistry and Pathophysiology: Change From Baseline to Week 48 in C-Telopeptide (CTX)
Description: CTX Week 48 difference from baseline
Time Frame: Baseline and wk 48
Population: Subjects with data for baseline and Week 48
Measure: Median (Full Range); unit: pM
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 70
pM | 25.90 [-819.51 to 1368.54]
Statistical Analysis 1: Comparison: Subjects Enrolled in ATN 110 or ATN 113; Test type: Other; p = 0.3483, Wilcoxon Signed Rank Test

63. Secondary Outcome: Change in Renal-endocrine-bone Biochemistry and Pathophysiology: Most Extreme Fold Change in Osteocalcin (OC)
Description: as for outcome 4
Time Frame: Baseline, Weeks 4, 8, 12, 24, 36 and 48
Population: Subjects with at least two measurements available for comparison
Measure: Median (Full Range); unit: fold change
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 90
fold change | 1.14 [0.67 to 1.76]

64. Secondary Outcome: Change in Renal-endocrine-bone Biochemistry and Pathophysiology: Most Extreme Fold Change in C-telopeptide (CTX)
Description: as for outcome 4
Time Frame: Baseline, Weeks 4, 8, 12, 24, 36 and 48
Population: Subjects with at least two measurements available for comparison
Measure: Median (Full Range); unit: fold change
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 90
fold change | 1.37 [0.74 to 4.05]

65. Secondary Outcome: Change in Renal-endocrine-bone Biochemistry and Pathophysiology: OC, Time to Most Extreme Fold Change
Description: as for outcome 5
Time Frame: Baseline, Weeks 4, 8, 12, 24, 36, and 48
Population: Subjects with at least two measurements available for comparison
Measure: Median (Full Range); unit: weeks
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 90
weeks | 12.00 [4.00 to 48.00]

66. Secondary Outcome: Change in Renal-endocrine-bone Biochemistry and Pathophysiology: Time to Most Extreme Fold Change in C-telopeptide (CTX)
Description: as for outcome 5
Time Frame: Baseline, Weeks 4, 8, 12, 24, 36, and 48
Population: Subjects with at least two measurements available for comparison
Measure: Median (Full Range); unit: weeks
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 90
weeks | 12.00 [4.00 to 48.00]

67. Secondary Outcome: Change in Renal-endocrine-bone Biochemistry and Pathophysiology: Slope of the Curve of Baseline to Most Extreme Fold Change in OC
Description: as for outcome 21
Time Frame: Baseline, Weeks 4, 8, 12, 24, 36, and 48
Population: Subjects with at least two measurements available for comparison
Measure: Median (Full Range); unit: (mcg/L)/ weeks
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 90
(mcg/L)/ weeks | 0.07 [-0.46 to 1.19]

68. Secondary Outcome: Change in Renal-endocrine-bone Biochemistry and Pathophysiology: Slope of the Curve of Baseline to Most Extreme Fold Change in CTX
Description: as for outcome 21
Time Frame: Baseline, Weeks (wks) 4, 8, 12, 24, 36, and 48
Population: Subjects with at least two measurements available for comparison
Measure: Median (Full Range); unit: (pM)/ weeks
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 90
(pM)/ weeks | 17.98 [-64.74 to 375.51]

69. Secondary Outcome: Area Under the Drug Concentration by Time Curve (AUC): Change From Baseline to Week 48 in PTH, by Overall Drug Exposure
Description: Overall drug exposure categories were determined based on the overall tertiles of mean AUC dried blood spot (DBS) Red Blood Cell (RBC) Tenofovir Diphosphate (intracellular) (TFV-DP). Comparisons were performed between the high exposure group and the low exposure group.
  The time points at which data were collected were: weeks 4, 8, 12, 24, 36, and 48.
Time Frame: Baseline and wk 48
Measure: Median (Full Range); unit: pg*wks/mL
Groups:
- High Exposure Group: Highest tertile of drug exposure, as measured by AUC (over the study duration) DBS RBC TFV-DP.
- Low Exposure Group: Lowest tertile of drug exposure, as measured by AUC (over the study duration) DBS RBC TFV-DP.
Arm/Group | High Exposure Group | Low Exposure Group
Number analyzed (Participants) | 23 | 19
pg*wks/mL | -0.09 [-16.18 to 26.87] | 3.59 [-13.39 to 24.54]
Statistical Analysis 1: Comparison: High Exposure Group vs Low Exposure Group; Test type: Other; p = 0.4043, Wilcoxon (Mann-Whitney)

70. Secondary Outcome: Area Under the Drug Concentration by Time Curve (AUC): Change From Baseline to Week 24 in PTH, by Overall Drug Exposure
Description: Overall drug exposure categories were determined based on the overall tertiles of mean AUC dried blood spot (DBS) Red Blood Cell (RBC) Tenofovir Diphosphate (intracellular) (TFV-DP). Comparisons were performed between the high exposure group and the low exposure group.
  The time points at which data were collected were: weeks 4, 8, 12, and 24.
Time Frame: Baseline and wk 24
Measure: Median (Full Range); unit: pg*wks/mL
Arm/Group | High Exposure Group | Low Exposure Group
Number analyzed (Participants) | 26 | 26
pg*wks/mL | 0.46 [-15.21 to 32.73] | 0.47 [-28.89 to 17.50]
Statistical Analysis 1: Comparison: High Exposure Group vs Low Exposure Group; Test type: Other; p = 0.2927, Wilcoxon (Mann-Whitney)

71. Secondary Outcome: Area Under the Drug Concentration by Time Curve (AUC): Change From Baseline to Week 24 in FGF23, by Overall Drug Exposure
Description: as for outcome 70
Time Frame: Baseline and wk 24
Measure: Median (Full Range); unit: pg*wks/mL
Arm/Group | High Exposure Group | Low Exposure Group
Number analyzed (Participants) | 26 | 26
pg*wks/mL | -6.88 [-27.23 to 17.18] | 0.79 [-62.55 to 26.42]
Statistical Analysis 1: Comparison: High Exposure Group vs Low Exposure Group; Test type: Other; p = 0.1134, Wilcoxon (Mann-Whitney)

72. Secondary Outcome: Area Under the Drug Concentration by Time Curve (AUC): Change From Baseline to Week 48 in FGF23, by Overall Drug Exposure
Description: as for outcome 69
Time Frame: Baseline and wk 48
Measure: Median (Full Range); unit: pg*wks/mL
Arm/Group | High Exposure Group | Low Exposure Group
Number analyzed (Participants) | 23 | 19
pg*wks/mL | 1.66 [-23.96 to 29.5] | 0.60 [-23.57 to 24.39]
Statistical Analysis 1: Comparison: High Exposure Group vs Low Exposure Group; Test type: Other; p = 0.5782, Wilcoxon (Mann-Whitney)

73. Secondary Outcome: Area Under the Drug Concentration by Time Curve (AUC): Change From Baseline to Week 24 in 1,25 OHD, by Overall Drug Exposure
Description: as for outcome 70
Time Frame: Baseline and wk 24
Measure: Median (Full Range); unit: pmol*wks/L
Arm/Group | High Exposure Group | Low Exposure Group
Number analyzed (Participants) | 27 | 26
pmol*wks/L | 10.80 [-117.15 to 91.65] | 7.07 [-123.12 to 228.28]
Statistical Analysis 1: Comparison: High Exposure Group vs Low Exposure Group; Test type: Other; p = 0.8658, Wilcoxon (Mann-Whitney)

74. Secondary Outcome: Area Under the Drug Concentration by Time Curve (AUC): Change From Baseline to Week 48 in 1,25 OHD, by Overall Drug Exposure
Description: as for outcome 69
Time Frame: Baseline and wk 48
Measure: Median (Full Range); unit: pmol*wks/L
Arm/Group | High Exposure Group | Low Exposure Group
Number analyzed (Participants) | 24 | 19
pmol*wks/L | -12.55 [-135.40 to 67.17] | -8.60 [-63.87 to 197.62]
Statistical Analysis 1: Comparison: High Exposure Group vs Low Exposure Group; Test type: Other; p = 0.5491, Wilcoxon (Mann-Whitney)

75. Secondary Outcome: Area Under the Drug Concentration by Time Curve (AUC): Change From Baseline to Week 24 in Osteocalcin (OC), by Overall Drug Exposure
Description: as for outcome 70
Time Frame: Baseline and wk 24
Measure: Median (Full Range); unit: mcg*wks/L
Arm/Group | High Exposure Group | Low Exposure Group
Number analyzed (Participants) | 26 | 26
mcg*wks/L | 0.87 [-3.61 to 4.63] | -1.03 [-4.87 to 5.02]
Statistical Analysis 1: Comparison: High Exposure Group vs Low Exposure Group; Test type: Other; p = 0.0238, Wilcoxon (Mann-Whitney)

76. Secondary Outcome: Area Under the Drug Concentration by Time Curve (AUC): Change From Baseline to Week 48 in Osteocalcin (OC), by Overall Drug Exposure
Description: as for outcome 69
Time Frame: Baseline and wk 48
Measure: Median (Full Range); unit: mcg*wks/L
Arm/Group | High Exposure Group | Low Exposure Group
Number analyzed (Participants) | 23 | 19
mcg*wks/L | 1.12 [-4.12 to 7.77] | -0.10 [-6.17 to 3.22]
Statistical Analysis 1: Comparison: High Exposure Group vs Low Exposure Group; Test type: Other; p = 0.1172, Wilcoxon (Mann-Whitney)

77. Secondary Outcome: Area Under the Drug Concentration by Time Curve (AUC): Change From Baseline to Week 24 in CTX, by Overall Drug Exposure
Description: as for outcome 70
Time Frame: Baseline and wk 24
Measure: Median (Full Range); unit: pM*wks
Arm/Group | High Exposure Group | Low Exposure Group
Number analyzed (Participants) | 26 | 26
pM*wks | 105.89 [-527.16 to 817.21] | -25.90 [-819.51 to 969.14]
Statistical Analysis 1: Comparison: High Exposure Group vs Low Exposure Group; Test type: Other; p = 0.1220, Wilcoxon (Mann-Whitney)

78. Secondary Outcome: Area Under the Drug Concentration by Time Curve (AUC): Change From Baseline to Week 48 in CTX, by Overall Drug Exposure
Description: as for outcome 69
Time Frame: Baseline and wk 48
Measure: Median (Full Range); unit: pM*wks
Arm/Group | High Exposure Group | Low Exposure Group
Number analyzed (Participants) | 23 | 19
pM*wks | 50.64 [-646.29 to 622.69] | -20.72 [-819.51 to 576.65]
Statistical Analysis 1: Comparison: High Exposure Group vs Low Exposure Group; Test type: Other; p = 1.000, Wilcoxon (Mann-Whitney)

79. Secondary Outcome: Area Under the Drug Concentration by Time Curve (AUC): Change From Baseline to Week 24 in SCr, by Overall Drug Exposure
Description: as for outcome 70
Time Frame: Baseline and wk 24
Measure: Median (Full Range); unit: mg*wks/dL
Arm/Group | High Exposure Group | Low Exposure Group
Number analyzed (Participants) | 27 | 26
mg*wks/dL | 0.02 [-0.09 to 0.14] | 0.00 [-0.19 to 0.13]

80. Secondary Outcome: Area Under the Drug Concentration by Time Curve (AUC): Change From Baseline to Week 48 in SCr, by Overall Drug Exposure
Description: as for outcome 69
Time Frame: Baseline and wk 48
Measure: Median (Full Range); unit: mg*wks/dL
Arm/Group | High Exposure Group | Low Exposure Group
Number analyzed (Participants) | 24 | 19
mg*wks/dL | 0.01 [-0.12 to 0.15] | -0.02 [-0.10 to 0.27]
Statistical Analysis 1: Comparison: High Exposure Group vs Low Exposure Group; Test type: Other; p = 0.7785, Wilcoxon (Mann-Whitney)

81. Secondary Outcome: Area Under the Drug Concentration by Time Curve (AUC): Change From Baseline to Week 24 in TRP, by Overall Drug Exposure
Description: as for outcome 70
Time Frame: Baseline and wk 24
Measure: Median (Full Range); unit: % of phosphorus reabsorbed*wks
Arm/Group | High Exposure Group | Low Exposure Group
Number analyzed (Participants) | 27 | 26
% of phosphorus reabsorbed*wks | 0.57 [-13.44 to 15.72] | 1.14 [-8.58 to 11.38]
Statistical Analysis 1: Comparison: High Exposure Group vs Low Exposure Group; Test type: Other; p = 0.4933, Wilcoxon (Mann-Whitney)

82. Secondary Outcome: Area Under the Drug Concentration by Time Curve (AUC): Change From Baseline to Week 48 in TRP, by Overall Drug Exposure
Description: as for outcome 69
Time Frame: Baseline and wk 48
Measure: Median (Full Range); unit: % of phosphorus reabsorbed*wks
Arm/Group | High Exposure Group | Low Exposure Group
Number analyzed (Participants) | 24 | 19
% of phosphorus reabsorbed*wks | 0.03 [-7.37 to 9.51] | -1.28 [-10.43 to 5.87]
Statistical Analysis 1: Comparison: High Exposure Group vs Low Exposure Group; Test type: Other; p = 0.5491, Wilcoxon (Mann-Whitney)

83. Secondary Outcome: Area Under the Drug Concentration by Time Curve (AUC): Change From Baseline to Week 24 in UCa/UCr Ratio, by Overall Drug Exposure
Description: as for outcome 70
Time Frame: Baseline and wk 24
Measure: Median (Full Range); unit: ratio*weeks
Arm/Group | High Exposure Group | Low Exposure Group
Number analyzed (Participants) | 27 | 26
ratio*weeks | 0.00 [-0.06 to 0.12] | -0.01 [-0.15 to 0.27]
Statistical Analysis 1: Comparison: High Exposure Group vs Low Exposure Group; Test type: Other; p = 0.5161, Wilcoxon (Mann-Whitney)

84. Secondary Outcome: Area Under the Drug Concentration by Time Curve (AUC): Change From Baseline to Week 48 in UCa/UCr Ratio, by Overall Drug Exposure
Description: as for outcome 69
Time Frame: Baseline and wk 48
Measure: Median (Full Range); unit: ratio*weeks
Arm/Group | High Exposure Group | Low Exposure Group
Number analyzed (Participants) | 24 | 19
ratio*weeks | 0.00 [-0.06 to 0.30] | 0.00 [-0.17 to 0.11]
Statistical Analysis 1: Comparison: High Exposure Group vs Low Exposure Group; Test type: Other; p = 0.5990, Wilcoxon (Mann-Whitney)

85. Secondary Outcome: Area Under the Drug Concentration by Time Curve (AUC): Change From Baseline to Week 24 in UB2MG, by Overall Drug Exposure
Description: as for outcome 70
Time Frame: Baseline and wk 24
Measure: Median (Full Range); unit: ng*wks/mL
Arm/Group | High Exposure Group | Low Exposure Group
Number analyzed (Participants) | 26 | 25
ng*wks/mL | -7.28 [-852.86 to 980.03] | -23.29 [-3716.53 to 1987.72]
Statistical Analysis 1: Comparison: High Exposure Group vs Low Exposure Group; Test type: Other; p = 0.8579, Wilcoxon (Mann-Whitney)

86. Secondary Outcome: Area Under the Drug Concentration by Time Curve (AUC): Change From Baseline to Week 48 in UB2MG, by Overall Drug Exposure
Description: as for outcome 69
Time Frame: Baseline and wk 48
Measure: Median (Full Range); unit: ng*wks/mL
Arm/Group | High Exposure Group | Low Exposure Group
Number analyzed (Participants) | 23 | 18
ng*wks/mL | -0.21 [-802.31 to 594.44] | -79.82 [-1152.17 to 393.80]
Statistical Analysis 1: Comparison: High Exposure Group vs Low Exposure Group; Test type: Other; p = 0.0719, Wilcoxon (Mann-Whitney)

87. Secondary Outcome: Area Under the Drug Concentration by Time Curve (AUC): Change From Baseline to Week 24 in UGluc, by Overall Drug Exposure
Description: as for outcome 70
Time Frame: Baseline and wk 24
Measure: Median (Full Range); unit: mg*wks/dL
Arm/Group | High Exposure Group | Low Exposure Group
Number analyzed (Participants) | 27 | 26
mg*wks/dL | -0.02 [-0.07 to 0.10] | 0.01 [-0.07 to 0.18]
Statistical Analysis 1: Comparison: High Exposure Group vs Low Exposure Group; Test type: Other; p = 0.3148, Wilcoxon (Mann-Whitney)

88. Secondary Outcome: Area Under the Drug Concentration by Time Curve (AUC): Change From Baseline to Week 48 in UGluc, by Overall Drug Exposure
Description: as for outcome 69
Time Frame: Baseline and wk 48
Measure: Median (Full Range); unit: mg*wks/dL
Arm/Group | High Exposure Group | Low Exposure Group
Number analyzed (Participants) | 24 | 19
mg*wks/dL | -0.01 [-0.09 to 0.06] | 0.02 [-0.09 to 0.10]
Statistical Analysis 1: Comparison: High Exposure Group vs Low Exposure Group; Test type: Other; p = 0.1390, Wilcoxon (Mann-Whitney)

89. Secondary Outcome: Area Under the Drug Concentration by Time Curve (AUC): Change From Baseline to Week 24 in URBP/UCr Ratio, by Overall Drug Exposure
Description: as for outcome 70
Time Frame: Baseline and wk 24
Measure: Median (Full Range); unit: mcg*wks/g
Arm/Group | High Exposure Group | Low Exposure Group
Number analyzed (Participants) | 26 | 24
mcg*wks/g | -2281.71 [-20957.98 to 23305.58] | 808.53 [-21627.73 to 11630.96]
Statistical Analysis 1: Comparison: High Exposure Group vs Low Exposure Group; Test type: Other; p = 0.2726, Wilcoxon (Mann-Whitney)

90. Secondary Outcome: Area Under the Drug Concentration by Time Curve (AUC): Change From Baseline to Week 48 in URBP/UCr Ratio, by Overall Drug Exposure
Description: as for outcome 69
Time Frame: Baseline and wk 48
Measure: Median (Full Range); unit: mcg*wks/g
Arm/Group | High Exposure Group | Low Exposure Group
Number analyzed (Participants) | 23 | 18
mcg*wks/g | -710.86 [-25872.11 to 12990.80] | 1606.38 [-29433.03 to 8572.38]
Statistical Analysis 1: Comparison: High Exposure Group vs Low Exposure Group; Test type: Other; p = 0.5370, Wilcoxon (Mann-Whitney)

91. Secondary Outcome: Area Under the Drug Concentration by Time Curve (AUC): Percent Change From Baseline to Week 24 in Lumbar Spine BMD, by Overall Drug Exposure
Description: as for outcome 70
Time Frame: Baseline and wk 24
Measure: Median (Full Range); unit: % change*wks
Arm/Group | High Exposure Group | Low Exposure Group
Number analyzed (Participants) | 26 | 26
% change*wks | -0.33 [-4.62 to 4.63] | 0.00 [-2.83 to 5.75]
Statistical Analysis 1: Comparison: High Exposure Group vs Low Exposure Group; Test type: Other; p = 0.2926, Wilcoxon (Mann-Whitney)

92. Secondary Outcome: Area Under the Drug Concentration by Time Curve (AUC): Percent Change From Baseline to Week 48 in Lumbar Spine BMD, by Overall Drug Exposure
Description: as for outcome 69
Time Frame: Baseline and wk 48
Measure: Median (Full Range); unit: % change*wks
Arm/Group | High Exposure Group | Low Exposure Group
Number analyzed (Participants) | 24 | 18
% change*wks | -0.32 [-4.47 to 3.74] | 0.88 [-2.44 to 7.98]
Statistical Analysis 1: Comparison: High Exposure Group vs Low Exposure Group; Test type: Other; p = 0.1906, Wilcoxon (Mann-Whitney)

93. Secondary Outcome: Area Under the Drug Concentration by Time Curve (AUC): Change From Baseline to Week 24 in Lumbar Spine BMD Z-score, by Overall Drug Exposure
Description: Overall drug exposure categories were determined based on the overall tertiles of mean AUC dried blood spot (DBS) Red Blood Cell (RBC) Tenofovir Diphosphate (intracellular) (TFV-DP). Comparisons were performed between the high exposure group and the low exposure group.
  The Z-score is the standard deviation around mean bone mineral density, adjusted for sex, age, and race/ethnicity. An average Z-score of zero would be expected in this group of healthy adolescents and young adults. An increase in Z-score would signify acceleration of accrual of bone mass, a positive outcome; a decrease in Z-score would signify either bone loss or failure to accrue the expected amount of bone mass, both of which are adverse outcomes. The Z-score is a normalized measure.
  The time points at which data were collected were: weeks 4, 8, 12, and 24.
Time Frame: Baseline and wk 24
Measure: Median (Full Range); unit: z-score
Arm/Group | High Exposure Group | Low Exposure Group
Number analyzed (Participants) | 26 | 26
z-score | -0.10 [-0.60 to 0.30] | 0.00 [-0.50 to 0.60]
Statistical Analysis 1: Comparison: High Exposure Group vs Low Exposure Group; Test type: Other; p = 0.2255, Wilcoxon (Mann-Whitney)

94. Secondary Outcome: Area Under the Drug Concentration by Time Curve (AUC): Change From Baseline to Week 48 in Lumbar Spine BMD Z-score, by Overall Drug Exposure
Description: Overall drug exposure categories were determined based on the overall tertiles of mean AUC dried blood spot (DBS) Red Blood Cell (RBC) Tenofovir Diphosphate (intracellular) (TFV-DP). Comparisons were performed between the high exposure group and the low exposure group.
  The Z-score is the standard deviation around mean bone mineral density, adjusted for sex, age, and race/ethnicity. An average Z-score of zero would be expected in this group of healthy adolescents and young adults. An increase in Z-score would signify acceleration of accrual of bone mass, a positive outcome; a decrease in Z-score would signify either bone loss or failure to accrue the expected amount of bone mass, both of which are adverse outcomes. The Z-score is a normalized measure.
  The time points at which data were collected were: weeks 4, 8, 12, 24, 36, and 48.
Time Frame: Baseline and wk 48
Measure: Median (Full Range); unit: z-score
Arm/Group | High Exposure Group | Low Exposure Group
Number analyzed (Participants) | 24 | 18
z-score | -0.20 [-0.50 to 0.20] | -0.10 [-0.80 to 0.60]
Statistical Analysis 1: Comparison: High Exposure Group vs Low Exposure Group; Test type: Other; p = 0.6285, Wilcoxon (Mann-Whitney)

95. Secondary Outcome: Area Under the Drug Concentration by Time Curve (AUC): Percent Change From Baseline to Week 24 in Femoral Neck BMD, by Overall Drug Exposure
Description: as for outcome 70
Time Frame: Baseline and wk 24
Measure: Median (Full Range); unit: % change*wks
Arm/Group | High Exposure Group | Low Exposure Group
Number analyzed (Participants) | 26 | 24
% change*wks | -0.80 [-7.34 to 2.31] | 0.62 [-3.89 to 8.13]
Statistical Analysis 1: Comparison: High Exposure Group vs Low Exposure Group; Test type: Other; p = 0.0148, Wilcoxon (Mann-Whitney)

96. Secondary Outcome: Area Under the Drug Concentration by Time Curve (AUC): Percent Change From Baseline to Week 48 in Femoral Neck BMD, by Overall Drug Exposure
Description: as for outcome 69
Time Frame: Baseline and wk 48
Measure: Median (Full Range); unit: % change*wks
Arm/Group | High Exposure Group | Low Exposure Group
Number analyzed (Participants) | 24 | 17
% change*wks | -1.89 [-5.09 to 4.39] | 1.14 [-2.54 to 8.48]
Statistical Analysis 1: Comparison: High Exposure Group vs Low Exposure Group; Test type: Other; p = 0.0166, Wilcoxon (Mann-Whitney)

97. Secondary Outcome: Area Under the Drug Concentration by Time Curve (AUC): Change From Baseline to Week 24 in Femoral Neck BMD Z-score, by Overall Drug Exposure
Description: as for outcome 93
Time Frame: Baseline and wk 24
Measure: Median (Full Range); unit: z-score
Arm/Group | High Exposure Group | Low Exposure Group
Number analyzed (Participants) | 25 | 24
z-score | -0.10 [-0.60 to 0.20] | 0.00 [-0.40 to 0.40]
Statistical Analysis 1: Comparison: High Exposure Group vs Low Exposure Group; Test type: Other; p = 0.0277, Wilcoxon (Mann-Whitney)

98. Secondary Outcome: Area Under the Drug Concentration by Time Curve (AUC): Change From Baseline to Week 48 in Femoral Neck BMD Z-score, by Overall Drug Exposure
Description: as for outcome 94
Time Frame: Baseline and wk 48
Measure: Median (Full Range); unit: z-score
Arm/Group | High Exposure Group | Low Exposure Group
Number analyzed (Participants) | 23 | 17
z-score | -0.10 [-0.50 to 0.30] | 0.10 [-0.70 to 0.40]
Statistical Analysis 1: Comparison: High Exposure Group vs Low Exposure Group; Test type: Other; p = 0.2610, Wilcoxon (Mann-Whitney)

99. Secondary Outcome: Area Under the Drug Concentration by Time Curve (AUC): Percent Change From Baseline to Week 24 in Total Body BMC, by Overall Drug Exposure
Description: as for outcome 70
Time Frame: Baseline and wk 24
Measure: Median (Full Range); unit: % change*wks
Arm/Group | High Exposure Group | Low Exposure Group
Number analyzed (Participants) | 26 | 26
% change*wks | -0.40 [-5.38 to 2.44] | -0.24 [-3.49 to 8.79]
Statistical Analysis 1: Comparison: High Exposure Group vs Low Exposure Group; Test type: Other; p = 0.4154, Wilcoxon (Mann-Whitney)

100. Secondary Outcome: Area Under the Drug Concentration by Time Curve (AUC): Percent Change From Baseline to Week 48 in Total Body BMC, by Overall Drug Exposure
Description: as for outcome 69
Time Frame: Baseline and wk 48
Measure: Median (Full Range); unit: % change*wks
Arm/Group | High Exposure Group | Low Exposure Group
Number analyzed (Participants) | 24 | 18
% change*wks | -0.60 [-7.69 to 3.08] | -1.24 [-3.79 to 12.21]
Statistical Analysis 1: Comparison: High Exposure Group vs Low Exposure Group; Test type: Other; p = 0.7125, Wilcoxon (Mann-Whitney)

101. Secondary Outcome: Magnitude of Change in Lumbar Spine BMD at Week 48
Description: The magnitude of change will be measured between Baseline and Week 48. For any given variable, at a given time point, the magnitude of change is the fold change compared to the baseline value (if multiplied by 100 would be the percent change from baseline).
Time Frame: Baseline and wk 48
Population: Subjects with data for Baseline and Week 48
Measure: Median (Full Range); unit: fold change
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 70
fold change | 1.00 [0.94 to 1.08]

102. Secondary Outcome: Magnitude of Change in Lumbar Spine BMD Z-score at Week 48
Description: The magnitude of change will be measured between Baseline and Week 48. For any given variable, at a given time point, the magnitude of change is the fold change compared to the baseline value (if multiplied by 100 would be the percent change from baseline).
  The Z-score is the standard deviation around mean bone mineral density, adjusted for sex, age, and race/ethnicity. An average Z-score of zero would be expected in this group of healthy adolescents and young adults. An increase in Z-score would signify acceleration of accrual of bone mass, a positive outcome; a decrease in Z-score would signify either bone loss or failure to accrue the expected amount of bone mass, both of which are adverse outcomes. The Z-score is a normalized measure.
Time Frame: Baseline and wk 48
Population: Subjects with data for Baseline and Week 48
Measure: Median (Full Range); unit: fold change
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 68
fold change | 1.04 [-0.33 to 4.50]

103. Secondary Outcome: Magnitude of Change in Femoral Neck BMD at Week 48
Description: as for outcome 101
Time Frame: Baseline and wk 48
Population: Subjects with data for Baseline and Week 48
Measure: Median (Full Range); unit: fold change
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 69
fold change | 1.00 [0.92 to 1.08]

104. Secondary Outcome: Magnitude of Change in Femoral Neck BMD Z-score at Week 48
Description: as for outcome 101
Time Frame: Baseline and wk 48
Population: Subjects with data for Baseline and Week 48
Measure: Median (Full Range); unit: fold change
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 62
fold change | 1.00 [-1.00 to 2.50]

105. Secondary Outcome: Magnitude of Change in Total Body BMC at Week 48
Description: as for outcome 101
Time Frame: Baseline and wk 48
Population: Subjects with data for Baseline and Week 48
Measure: Median (Full Range); unit: fold change
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 70
fold change | 1.00 [0.92 to 1.12]

106. Secondary Outcome: Changes in BMD/BMC in the Extension Phase: Lumbar Spine BMD Change at EPH1 From Baseline
Description: For subjects in the extension phase of the study, the last measured values at the ATN 110 or ATN 113 study week 48 visit will be compared with those measured at the Extension Phase visit 1 (EPH 1, 24 weeks after the ATN 110 or ATN 113 study week 48 visit) and EPH 2 (48 weeks after the ATN 110 or ATN 113 study week 48 visit).
  This measure shows the difference between the Baseline measure and the first Extension Phase visit (BL - EPH1)
Time Frame: Baseline and wk 72
Population: Subjects who meet specific bone or renal criteria at Week 48 of the ATN 110 or ATN 113 study will be followed for an additional 48 weeks in the Extension Phase.
Measure: Median (Full Range); unit: g/cm^2
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 37
g/cm^2 | -0.01 [-0.067 to 0.056]

107. Secondary Outcome: Changes in BMD/BMC in the Extension Phase: Lumbar Spine BMD Change at EPH2 From Baseline
Description: For subjects in the extension phase of the study, the last measured values at the ATN 110 or ATN 113 study week 48 visit will be compared with those measured at the Extension Phase visit 1 (EPH 1, 24 weeks after the ATN 110 or ATN 113 study week 48 visit) and EPH 2 (48 weeks after the ATN 110 or ATN 113 study week 48 visit).
  This measure shows the difference between the Baseline measure and the second Extension Phase visit (BL - EPH2)
Time Frame: Baseline and wk 96
Population: as for outcome 106
Measure: Median (Full Range); unit: g/cm^2
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 40
g/cm^2 | -0.01 [-0.07 to 0.06]

108. Secondary Outcome: Changes in BMD/BMC in the Extension Phase: Lumbar Spine BMD Change at EPH1 From Week 48 (or Last Visit on Study)
Description: For subjects in the extension phase of the study, the last measured values at the ATN 110 or ATN 113 study week 48 visit will be compared with those measured at the Extension Phase visit 1 (EPH 1, 24 weeks after the ATN 110 or ATN 113 study week 48 visit) and EPH 2 (48 weeks after the ATN 110 or ATN 113 study week 48 visit).
  This measure shows the difference between the last measure on study and the first Extension Phase visit (Last - EPH1)
Time Frame: Wk 48 (or last available measurement on study), Wk 72
Population: as for outcome 106
Measure: Median (Full Range); unit: g/cm^2
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 37
g/cm^2 | -0.01 [-0.07 to 0.03]

109. Secondary Outcome: Changes in BMD/BMC in the Extension Phase: Lumbar Spine BMD Change at EPH2 From Week 48 (or Last Visit on Study)
Description: For subjects in the extension phase of the study, the last measured values at the ATN 110 or ATN 113 study week 48 visit will be compared with those measured at the Extension Phase visit 1 (EPH 1, 24 weeks after the ATN 110 or ATN 113 study week 48 visit) and EPH 2 (48 weeks after the ATN 110 or ATN 113 study week 48 visit).
  This measure shows the difference between the last measure on study and the second Extension Phase visit (Last - EPH2)
Time Frame: Wk 48 (or last available measurement on study), Wk 96
Population: as for outcome 106
Measure: Median (Full Range); unit: g/cm^2
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 40
g/cm^2 | -0.01 [-0.09 to 0.05]

110. Secondary Outcome: Changes in BMD/BMC in the Extension Phase: Lumbar Spine BMD Z-score Change at EPH1 From Baseline
Description: For subjects in the extension phase of the study, the last measured values at the ATN 110 or ATN 113 study week 48 visit will be compared with those measured at the Extension Phase visit 1 (EPH 1, 24 weeks after the ATN 110 or ATN 113 study week 48 visit) and EPH 2 (48 weeks after the ATN 110 or ATN 113 study week 48 visit).
  This measure shows the difference between the Baseline measure and the first Extension Phase visit (BL - EPH1).
  The Z-score is the standard deviation around mean bone mineral density, adjusted for sex, age, and race/ethnicity. An average Z-score of zero would be expected in this group of healthy adolescents and young adults. An increase in Z-score would signify acceleration of accrual of bone mass, a positive outcome; a decrease in Z-score would signify either bone loss or failure to accrue the expected amount of bone mass, both of which are adverse outcomes. The Z-score is a normalized measure.
Time Frame: Baseline and wk 72
Population: as for outcome 106
Measure: Median (Full Range); unit: z-score
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 37
z-score | 0.10 [-0.60 to 1.00]

111. Secondary Outcome: Changes in BMD/BMC in the Extension Phase: Lumbar Spine BMD Z-score Change at EPH2 From Baseline
Description: For subjects in the extension phase of the study, the last measured values at the ATN 110 or ATN 113 study week 48 visit will be compared with those measured at the Extension Phase visit 1 (EPH 1, 24 weeks after the ATN 110 or ATN 113 study week 48 visit) and EPH 2 (48 weeks after the ATN 110 or ATN 113 study week 48 visit).
  This measure shows the difference between the Baseline measure and the second Extension Phase visit (BL - EPH2)
  The Z-score is the standard deviation around mean bone mineral density, adjusted for sex, age, and race/ethnicity. An average Z-score of zero would be expected in this group of healthy adolescents and young adults. An increase in Z-score would signify acceleration of accrual of bone mass, a positive outcome; a decrease in Z-score would signify either bone loss or failure to accrue the expected amount of bone mass, both of which are adverse outcomes. The Z-score is a normalized measure.
Time Frame: Baseline and wk 96
Population: as for outcome 106
Measure: Median (Full Range); unit: z-score
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 40
z-score | 0.20 [-0.60 to 0.90]

112. Secondary Outcome: Changes in BMD/BMC in the Extension Phase: Lumbar Spine BMD Z-score Change at EPH1 From Week 48 (or Last Visit on Study)
Description: For subjects in the extension phase of the study, the last measured values at the ATN 110 or ATN 113 study week 48 visit will be compared with those measured at the Extension Phase visit 1 (EPH 1, 24 weeks after the ATN 110 or ATN 113 study week 48 visit) and EPH 2 (48 weeks after the ATN 110 or ATN 113 study week 48 visit).
  This measure shows the difference between the last measure on study and the first Extension Phase visit (Last - EPH1)
  The Z-score is the standard deviation around mean bone mineral density, adjusted for sex, age, and race/ethnicity. An average Z-score of zero would be expected in this group of healthy adolescents and young adults. An increase in Z-score would signify acceleration of accrual of bone mass, a positive outcome; a decrease in Z-score would signify either bone loss or failure to accrue the expected amount of bone mass, both of which are adverse outcomes. The Z-score is a normalized measure.
Time Frame: Wk 48 (or last available measurement on study), Wk 72
Population: as for outcome 106
Measure: Median (Full Range); unit: z-score
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 37
z-score | 0.00 [-0.50 to 0.30]

113. Secondary Outcome: Changes in BMD/BMC in the Extension Phase: Lumbar Spine BMD Z-score Change at EPH2 From Week 48 (or Last Visit on Study)
Description: For subjects in the extension phase of the study, the last measured values at the ATN 110 or ATN 113 study week 48 visit will be compared with those measured at the Extension Phase visit 1 (EPH 1, 24 weeks after the ATN 110 or ATN 113 study week 48 visit) and EPH 2 (48 weeks after the ATN 110 or ATN 113 study week 48 visit).
  This measure shows the difference between the last measure on study and the second Extension Phase visit (Last - EPH2)
  The Z-score is the standard deviation around mean bone mineral density, adjusted for sex, age, and race/ethnicity. An average Z-score of zero would be expected in this group of healthy adolescents and young adults. An increase in Z-score would signify acceleration of accrual of bone mass, a positive outcome; a decrease in Z-score would signify either bone loss or failure to accrue the expected amount of bone mass, both of which are adverse outcomes. The Z-score is a normalized measure.
Time Frame: Wk 48 (or last available measurement on study), Wk 96
Population: as for outcome 106
Measure: Median (Full Range); unit: z-score
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 40
z-score | 0.00 [-0.50 to 0.40]

114. Secondary Outcome: Changes in BMD/BMC in the Extension Phase: Femoral Neck BMD Change at EPH1 From Baseline
Description: as for outcome 106
Time Frame: Baseline and wk 72
Population: as for outcome 106
Measure: Median (Full Range); unit: g/cm^2
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 37
g/cm^2 | 0.01 [-0.06 to 0.05]

115. Secondary Outcome: Changes in BMD/BMC in the Extension Phase: Femoral Neck BMD Change at EPH2 From Baseline
Description: as for outcome 107
Time Frame: Baseline and wk 96
Population: as for outcome 106
Measure: Median (Full Range); unit: g/cm^2
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 40
g/cm^2 | 0.00 [-0.07 to 0.10]

116. Secondary Outcome: Changes in BMD/BMC in the Extension Phase: Femoral Neck BMD Change at EPH1 From Week 48 (or Last Visit on Study)
Description: For subjects in the extension phase of the study, the last measured values at the ATN 110 or ATN 113 study week 48 visit will be compared with those measured at the Extension Phase visit 1 (EPH 1, 24 weeks after the ATN 110 or ATN 113 study week 48 visit) and EPH 2 (48 weeks after the ATN 110 or ATN 113 study week 48 visit).
  This measure shows the difference between the last measure on study and the first Extension Phase visit (Last- EPH1)
Time Frame: Wk 48 (or last available measurement on study), Wk 72
Population: as for outcome 106
Measure: Median (Full Range); unit: g/cm^2
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 37
g/cm^2 | 0.00 [-0.06 to 0.09]

117. Secondary Outcome: Changes in BMD/BMC in the Extension Phase: Femoral Neck BMD Change at EPH2 From Week 48 (or Last Visit on Study)
Description: For subjects in the extension phase of the study, the last measured values at the ATN 110 or ATN 113 study week 48 visit will be compared with those measured at the Extension Phase visit 1 (EPH 1, 24 weeks after the ATN 110 or ATN 113 study week 48 visit) and EPH 2 (48 weeks after the ATN 110 or ATN 113 study week 48 visit).
  This measure shows the difference between the last measure on study and the second Extension Phase visit (Last- EPH2)
Time Frame: W 48 (or last available measurement on study), Wk 96
Population: as for outcome 106
Measure: Median (Full Range); unit: g/cm^2
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 40
g/cm^2 | -0.01 [-0.10 to 0.08]

118. Secondary Outcome: Changes in BMD/BMC in the Extension Phase: Femoral Neck BMD Z-score Change at EPH1 From Baseline
Description: For subjects in the extension phase of the study, the last measured values at the ATN 110 or ATN 113 study week 48 visit will be compared with those measured at the Extension Phase visit 1 (EPH 1, 24 weeks after the ATN 110 or ATN 113 study week 48 visit) and EPH 2 (48 weeks after the ATN 110 or ATN 113 study week 48 visit).
  This measure shows the difference between the Baseline measure and the first Extension Phase visit (BL - EPH1)
  The Z-score is the standard deviation around mean bone mineral density, adjusted for sex, age, and race/ethnicity. An average Z-score of zero would be expected in this group of healthy adolescents and young adults. An increase in Z-score would signify acceleration of accrual of bone mass, a positive outcome; a decrease in Z-score would signify either bone loss or failure to accrue the expected amount of bone mass, both of which are adverse outcomes. The Z-score is a normalized measure.
Time Frame: Baseline and wk 72
Population: as for outcome 106
Measure: Median (Full Range); unit: z-score
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 35
z-score | 0.10 [-0.30 to 0.70]

119. Secondary Outcome: Changes in BMD/BMC in the Extension Phase: Femoral Neck BMD Z-score Change at EPH2 From Baseline
Description: as for outcome 111
Time Frame: Baseline, Week 96
Population: as for outcome 106
Measure: Median (Full Range); unit: z-score
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 38
z-score | 0.10 [-0.50 to 0.80]

120. Secondary Outcome: Changes in BMD/BMC in the Extension Phase: Femoral Neck BMD Z-score Change at EPH1 From Week 48 (or Last Visit on Study)
Description: as for outcome 112
Time Frame: Week 48 (or last available measurement on study), Week 72
Population: as for outcome 106
Measure: Median (Full Range); unit: z-score
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 37
z-score | 0.00 [-0.40 to 0.70]

121. Secondary Outcome: Changes in BMD/BMC in the Extension Phase: Femoral Neck BMD Z-score Change at EPH2 From Week 48 (or Last Visit on Study)
Description: For subjects in the extension phase of the study, the last measured values at the ATN 110 or ATN 113 study week 48 visit will be compared with those measured at the Extension Phase visit 1 (EPH 1, 24 weeks after the ATN 110 or ATN 113 study week 48 visit) and EPH 2 (48 weeks after the ATN 110 or ATN 113 study week 48 visit).
  This measure shows the difference between the last measure on study and the second Extension Phase visit (Last - EPH2).
  The Z-score is the standard deviation around mean bone mineral density, adjusted for sex, age, and race/ethnicity. An average Z-score of zero would be expected in this group of healthy adolescents and young adults. An increase in Z-score would signify acceleration of accrual of bone mass, a positive outcome; a decrease in Z-score would signify either bone loss or failure to accrue the expected amount of bone mass, both of which are adverse outcomes. The Z-score is a normalized measure.
Time Frame: Wk 48 (or last available measurement on study), Wk 96
Population: as for outcome 106
Measure: Median (Full Range); unit: z-score
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 40
z-score | -0.05 [-0.60 to 0.60]

122. Secondary Outcome: Changes in BMD/BMC in the Extension Phase: Total Body BMC Change at EPH1 From Baseline
Description: as for outcome 106
Time Frame: Baseline and wk 72
Population: as for outcome 106
Measure: Median (Full Range); unit: g
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 37
g | 7.90 [-105.01 to 129.00]

123. Secondary Outcome: Changes in BMD/BMC in the Extension Phase: Total Body BMC Change at EPH2 From Baseline
Description: as for outcome 107
Time Frame: Baseline and wk 96
Population: as for outcome 106
Measure: Median (Full Range); unit: g
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 40
g | -17.49 [-275.00 to 93.65]

124. Secondary Outcome: Changes in BMD/BMC in the Extension Phase: Total Body BMC Change at EPH1 From Week 48 (or Last Visit on Study)
Description: as for outcome 116
Time Frame: Wk 48 (or last available measurement on study), Wk 72
Population: as for outcome 106
Measure: Median (Full Range); unit: g
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 37
g | -27.80 [-80.09 to 65.00]

125. Secondary Outcome: Changes in BMD/BMC in the Extension Phase: Total Body BMC Change at EPH2 From Week 48 (or Last Visit on Study)
Description: as for outcome 117
Time Frame: Wk 48 (or last available measurement on study), Wk 96
Population: as for outcome 106
Measure: Median (Full Range); unit: g
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Number analyzed (Participants) | 40
g | -46.83 [-145.00 to 41.84]

ADVERSE EVENTS:
Time Frame: Adverse Event data not collected through this study; see reporting description below.
Description: Serious and/or Other [Not Including Serious] Adverse Events were not monitored/assessed through this sub-study; instead, all monitoring of adverse events in ATN 117 (NCT01769469) subjects occurred through the ATN 110 (NCT01772823) or ATN 113 (NCT01769456) studies in which ATN 117 (NCT01769469) subjects were initially enrolled.
Arm/Group | Subjects Enrolled in ATN 110 or ATN 113
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Since high and low drug exposure groups were not assigned by the study team, but rather "chosen" by the participants and categorized post hoc for analysis, there may be unidentified variables confounding our findings.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Adolescent Medicine Trials Network (ATN) for HIV/AIDS Interventions Publication Policy outlines procedures for the development and review of abstracts, publications and presentations. The Adolescent Medicine Leadership Group (AMLG) retains custody of and primary rights to the data. Use of data must be approved by the protocol team and AMLG.